CLINICAL TRIAL: NCT03015129
Title: A Phase 2 Trial of Durvalumab [MEDI4736](Anti-PD-L1 Antibody) With or Without Tremelimumab (Anti-CTLA-4 Antibody) in Patients With Persistent or Recurrent Endometrial Carcinoma and Endometrial Carcinosarcoma
Brief Title: A Study of Durvalumab With or Without Tremelimumab in Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1491
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-01

CONDITIONS: Endometrial Cancer; Endometrial Carcinosarcoma; Endometrial Carcinoma; Endometrial Cancer Recurrent; Endometrial Carcinoma, Recurrent
Keywords: Durvalumab; MEDI4736; Tremelimumab; anti-PD-L1 Antibody; anti-CTLA-4 antibody; 16-1491
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Durvalubmab (Experimental): Patients will receive intravenous infusion of durvalumab 1500mg Fixed Dose every 4 weeks until patient develops a loss of clinical benefit or experiences unacceptable toxicities.
  Interventions: Drug: Durvalumab
- Durvalubmab + Tremelimumab (Experimental): Patients will receive 1500mg Flat Dose durvalubmab via intravenous infusion every 4 weeks for up to 4 cycles and 75mg tremelimumab via intravenous infusion every 4 weeks for up to 4 cycles, and then continue 1500mg Fixed Dose durvalumab every 4 weeks until patient develops a loss of clinical benefit or experiences unacceptable toxicities.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab
Drug: Tremelimumab
  Arms: Durvalubmab + Tremelimumab

SUMMARY:
This study will test the safety and efficacy of the experimental drug called durvalumab with or without another experimental drug called tremelimumab in endometrial cancer.

Radiologic tumor assessment will be repeated every 8 weeks +/- 7 days for the first 48 weeks and then every 12 weeks +/- 7 days until PD. For patients who remain progression free 2 years post completion of protocol directed treatment, every 6 months +/- 1 month. irRECIST assessments will only be completed for patients continuing treatment beyond PD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have recurrent or persistent endometrial carcinoma (including: Endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, dedifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell carcinoma, and transitional cell carcinoma) or endometrial carcinosarcoma). Histologic documentation of diagnosis of carcinoma is required. MSI-high patients will be identified based on immunohistochemistry or MSI testing of archival tumor specimens by department of pathology or via known mutations found in mismatch repair genes via the Integrated Mutation Profiling of Actionable Cancer Targets (IMPACT) assay through MSKCC IRB# 12-245.
* All patients must have measurable disease. Measurable disease is defined by RECIST (version 1.1). Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be ≥ 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or ≥ 20 mm when measured by chest x-ray. Lymph nodes must be ≥ 15 mm in short axis when measured by CT or MRI.
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST version 1.1. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
* Age ≥ 18 years and life expectancy of ≥ 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Resolution of (non-laboratory) adverse effects of recent surgery, radiotherapy, or chemotherapy to Grade ≤1 prior to first study treatment (with the exception of alopecia or neuropathy).
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of endometrial carcinoma or carcinosarcoma. Initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy. Chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen.
* Patients are allowed to receive, but are not required to receive, three additional cytotoxic regimen for management of recurrent or persistent disease. Hormonal therapies will not count toward the prior regimen limit.
* Adequate normal organ and marrow function defined by the following laboratory results obtained within 14 days prior to first treatment:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (> 1500 per mm^3)
  * Platelet ≥ 100 x 10^9/L (>100,000 per mm^3)
  * Hemoglobin ≥ 9.0 g/dL
  * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). (Unless Gilbert's Syndrome,for which Bilirubin ≤ 3 x institutional upper limit of normal (ULN) without concurrent clinically significant liver disease)
  * AST (SGOT)/ALT (SGPT) ≤ 3 x institutional upper limit of normal unless (ULN) unless liver metastases are present, in which case it must be ≤ 5x ULN
  * Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN)
* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥55 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Patients must have been enrolled, or agree to consent to the companion genomic profiling study MSKCC IRB# 12-245. Results must be available before starting treatment on protocol.
* Patients must have signed an approved informed consent and authorization permitting release of personal information.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site); Previous enrollment in the present study.
* Participation in another clinical study with receipt of an investigational product during the last 4 weeks
* Any previous treatment with a PD-1 or PD-L1 inhibitor, including durvalumab or any anti-CTLA4, including tremelimumab.
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease (eg, cervical cancer in situ)
  * Adequately treated stage 1 breast cancer.
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) < 21 days prior to the first dose of study drug. Receipt of the last dose of hormonal therapy within < 7 days prior to the first dose of study drug.
* Any prior radiation therapy must be discontinued at least four weeks prior to registration.
* At least 4 weeks must have elapsed since the patient underwent any major surgery (e.g., major: laparotomy, laparoscopy) There is no delay in treatment for minor procedures (e.g., central venous access catheter placement).
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs)
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or durvalumab and tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., dexamethasone for nausea or steroids as CT scan contrast premedication) may be enrolled.
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > Grade 1
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History and/or confirmed pneumonitis or interstitial lung disease
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab or any excipient
* History of hypersensitivity to tremelimumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.
* Subjects with uncontrolled seizures.
* Patients who are pregnant or breastfeeding or patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period
* History of small or large bowel obstruction within 3 months of registration, including subjects with palliative gastric drainage catheters. Subjects with palliative diverting ileostomy or colostomy are allowed if they have been symptom-free for more than 3 months.
* Ongoing bowel perforation or presence of bowel fistula or abscess within 3 months of registration.
* Subjects with refractory ascites, defined as ascites needing drainage catheter or therapeutic paracentesis more often than every 4 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01; Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Makker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Di Dio C, Bogani G, Di Donato V, Cuccu I, Muzii L, Musacchio L, Scambia G, Lorusso D. The role of immunotherapy in advanced and recurrent MMR deficient and proficient endometrial carcinoma. Gynecol Oncol. 2023 Feb;169:27-33. doi: 10.1016/j.ygyno.2022.11.031. Epub 2022 Dec 6. PMID 36493574
- [Derived] Antill Y, Kok PS, Robledo K, Yip S, Cummins M, Smith D, Spurdle A, Barnes E, Lee YC, Friedlander M, Baron-Hay S, Shannon C, Coward J, Beale P, Goss G, Meniawy T, Lombard J, Andrews J, Stockler MR, Mileshkin L; Australia New Zealand Gynaecological Oncology Group (ANZGOG). Clinical activity of durvalumab for patients with advanced mismatch repair-deficient and repair-proficient endometrial cancer. A nonrandomized phase 2 clinical trial. J Immunother Cancer. 2021 Jun;9(6):e002255. doi: 10.1136/jitc-2020-002255. PMID 34103352
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Durvalubmab: Patients will receive intravenous infusion of durvalumab 1500mg Fixed Dose every 4 weeks until patient develops a loss of clinical benefit or experiences unacceptable toxicities.
  Durvalumab
- Durvalubmab + Tremelimumab: Patients will receive 1500mg Flat Dose durvalubmab via intravenous infusion every 4 weeks for up to 4 cycles and 75mg tremelimumab via intravenous infusion every 4 weeks for up to 4 cycles, and then continue 1500mg Fixed Dose durvalumab every 4 weeks until patient develops a loss of clinical benefit or experiences unacceptable toxicities.
  Durvalumab
  Tremelimumab
Period: Overall Study
Arm/Group | Durvalubmab | Durvalubmab + Tremelimumab
Started | 40 | 40
Completed | 0 | 0
Not Completed | 40 | 40
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Progression of disease | 38 | 33
Not completed — Adverse Event | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalubmab | Durvalubmab + Tremelimumab | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Full Range); unit: years] | 65 [45 to 78] | 66 [52 to 84] | 66 [45 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 39 | 37 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 29 | 27 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Treatment Efficacy Determined by Measuring the Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 72 months
Measure: Number; unit: Participants
Arm/Group | Durvalubmab | Durvalubmab + Tremelimumab
Number analyzed (Participants) | 40 | 40
Participants | 5 | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Durvalubmab | Durvalubmab + Tremelimumab
All-Cause Mortality (participants affected / at risk) | 2/40 | 2/40
Serious Adverse Events (participants affected / at risk) | 13/40 | 7/40
Other Adverse Events (participants affected / at risk) | 39/40 | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalubmab (N=40) | Durvalubmab + Tremelimumab (N=40)
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Edema cerebral (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 2 | 2
Fever (General disorders) | 3 | 1
Hematoma (Vascular disorders) | 0 | 1
Hypercalcemia (General disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 6 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
CPK increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Muscle weakness left-sided (Nervous system disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Weight Loss (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalubmab (N=40) | Durvalubmab + Tremelimumab (N=40)
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 25 | 12
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Anal pain (Gastrointestinal disorders) | 3 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 12 | 5
Anxiety (Psychiatric disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 11
Ascites (Gastrointestinal disorders) | 2 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Bladder infection (Infections and infestations) | 4 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 3 | 0
Confusion (Psychiatric disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 12 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Creatinine Increased (Investigations) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 22 | 10
Dizziness (Nervous system disorders) | 4 | 9
Dry mouth (Gastrointestinal disorders) | 3 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Edema limbs (General disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 3
Fatigue (General disorders) | 26 | 20
Fever (General disorders) | 3 | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 3 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Gum infection (Infections and infestations) | 0 | 8
Headache (Nervous system disorders) | 3 | 0
Hematoma (Vascular disorders) | 0 | 2
Hot flashes (Vascular disorders) | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hypertension (Vascular disorders) | 14 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 0 | 4
Increased Urinary Frequency (Renal and urinary disorders) | 6 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3
Lymphedema (Vascular disorders) | 2 | 0
Memory impairment (Nervous system disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Nausea (Gastrointestinal disorders) | 11 | 15
Non-cardiac chest pain (General disorders) | 0 | 2
Pain (General disorders) | 17 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 11
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 6
Sinus bradycardia (Cardiac disorders) | 2 | 0
Sinusitis (Infections and infestations) | 0 | 2
Skin infection (Infections and infestations) | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 3 | 4
Upper respiratory infection (Infections and infestations) | 2 | 2
Urinary frequency (Renal and urinary disorders) | 3 | 2
Urinary hesitancy (Renal and urinary disorders) | 0 | 4
Urinary tract infection (Infections and infestations) | 8 | 4
Urinary tract pain (Renal and urinary disorders) | 3 | 7
Urinary urgency (Renal and urinary disorders) | 2 | 1
Vaginal discharge (Reproductive system and breast disorders) | 4 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 | 3
Vaginal yeast (Reproductive system and breast disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 10 | 6
Weight gain (Investigations) | 6 | 5
Weight loss (Investigations) | 16 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT03015129/Prot_SAP_000.pdf